CLINICAL TRIAL: NCT03391934
Title: A Phase III, Randomized, Two-armed, Parallel, Double-blind, Active-controlled, Equivalency Clinical Trial of Cetuximab (CinnaGen Co.) Efficacy and Safety Compared With Erbitux (Merck Co.) and FOLFIRI for RAS Wild-type mCRC
Brief Title: Comparing Efficacy and Safety of Cetuximab (CinnaGen) Versus Erbitux® (Merck) in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cinnagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CET.CIN.HR.96 (III)
Record Dates: First submitted 2017-12-31; First posted 2018-01-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: RAS Wild-type; Cetuximab; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Leucovorin; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both of the drugs used in the study are indistinguishable for patients and their respective curative staff because they are similar in size and shape of the vials, caps, aluminum sealing and paints, and it is not possible to distinguish the type of brand from the appearance of the vials. Additionally, people who are evaluating the results and analyzing data are not aware of the type of patient grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cetuximab+ FOLFIRI (Experimental): Cetuximab (Produced by CinnaGen Co.): 400 mg/m2 weekly in the first dose and 250 mg/m2 in the next doses Irinitecan: 180 mg/m2 biweekly Leucovorin: 400 mg/m2 biweekly Fluorouracil: 400 mg/m2 push, and 2400 mg/m2 as 46-h infusion biweekly
  Interventions: Drug: Cetuximab + FOLFIRI
- Cetuximab + FOLFIRI (Active Comparator): Erbitux® (Produced by Merk Co.): 400 mg/m2 weekly Irinitecan: 180 mg/m2 biweekly Leucovorin: 400 mg/m2 biweekly Fluorouracil: 400 mg/m2 push, and 2400 mg/m2 as 46-h infusion biweekly
  Interventions: Drug: Cetuximab + FOLFIRI

INTERVENTIONS:
Drug: Cetuximab + FOLFIRI — Cetuximab 400 mg/m2 will be administered in the first dose and 250 mg/m2 will be administered in the next doses every week. Irinotecan will be administered 180 mg/m2 biweekly. Leucovorin will be administered 400 mg/m2 biweekly.Fluorouracil will be administered 400 mg/m2 push, and 2400 mg/m2 as 46-h infusion biweekly.
  Other Names: FOLFIRI = irinotecan + calcium folinate + 5-fluorouracil

SUMMARY:
The study is designed as phase III, randomized, two armed, parallel, double blind (patient and assessor blinded), active controlled, and equivalency clinical trial with primary endpoint of Progression-Free Survival of Cetuximab® (produced by CinnaGen) compared with Erbitux® (Cetuximab, the reference drug) in patients with RAS wild-type Metastatic Colorectal Cancer with the allocation ratio of 2:1.Patients who met the following criteria could be recruited to receive the mentioned intervention randomly. Inclusion criteria: Male or female older than 18 years old, histologically confirmed adenocarcinoma of the colon or rectum which is metastatic, having one or more bi-dimensionally measurable lesions as defined by RECIST criteria, tumor that could not be resected for curative purposes,ECOG performance status score of 2 or less,life expectancy of longer than 3 months (clinical assessment),evidence of tumor EGFR expression (expanded wild-type RAS),adequate organ and marrow function as defined:

ANC ≥ 1,500/mm3 Plt ≥ 100,000/mm3 Hb ≥ 9 g/dL (may have had blood transfusions) AST/ALT ≤ 2.5 IULN or ≤ 5 IULN with known liver metastases Total bilirubin ≤ 1.5 IULN Serum Creatinine ≤ 1.5 IULN INR ≤ 1.5 and PTT ≤ 1.5 IULN

DETAILED DESCRIPTION:
The study is designed as phase III, randomized, two armed, parallel, double blind (patient and assessor blinded), active controlled, and equivalency clinical trial with primary endpoint of Progression-Free Survival of Cetuximab® (produced by CinnaGen) compared with Erbitux® (Cetuximab, the reference drug) in patients with RAS wild-type Metastatic Colorectal Cancer with the allocation ratio of 2:1.Patients who met the following criteria could be recruited to receive the mentioned intervention randomly. Inclusion criteria: Male or female older than 18 years old, histologically confirmed adenocarcinoma of the colon or rectum which is metastatic, having one or more bi-dimensionally measurable lesions as defined by RECIST criteria, tumor that could not be resected for curative purposes,ECOG performance status score of 2 or less,life expectancy of longer than 3 months (clinical assessment),evidence of tumor EGFR expression (expanded wild-type RAS),adequate organ and marrow function as defined:

ANC ≥ 1,500/mm3 Plt ≥ 100,000/mm3 Hb ≥ 9 g/dL (may have had blood transfusions) AST/ALT ≤ 2.5 IULN or ≤ 5 IULN with known liver metastases Total bilirubin ≤ 1.5 IULN Serum Creatinine ≤ 1.5 IULN INR ≤ 1.5 and PTT ≤ 1.5 IULN

Patients who have previous exposure to an anti-EGFR therapy or irinotecan-based chemotherapy, radiotherapy, surgery (excluding previous diagnostic biopsy), or any investigational drug in the 30-day period before the start of treatment in our trial will be excluded from the study. Also, female patients who are pregnant or lactating, and patients with any history of another primary malignancy in the past five years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix, and patients with inability to comply with the study and/or follow up procedures will be excluded.The primary endpoint of the study is Progression-Free Survival (PFS) defined as the time from randomization to disease progression or death from any cause. The secondary endpoints of the study are Overall Survival (OS) defined as the time from date of randomization to date of death due to any cause, Objective Response Rate (ORR) defined as the sum of partial and complete responses, according to RECIST criteria and Time to Treatment Failure (TTF) is defined as the time from the date of randomization to the date of each of the following:

The treatment modalities did not destroy or modify the cancer cells, The tumor either became larger (disease progression) or stayed the same size after treatment, Discontinuation of treatment, Death from any cause

Safety and Immunogenicity will also be assessed during the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 18 years old
* Histologically confirmed adenocarcinoma of the colon or rectum which is metastatic
* Having one or more bi-dimensionally measurable lesions as defined by RECIST criteria
* Tumor that could not be resected for curative purposes
* ECOG performance status score of 2 or less
* Life expectancy of longer than 3 months (clinical assessment)
* Evidence of tumor EGFR expression (expanded wild-type RAS)
* Adequate organ and marrow function as defined:

ANC ≥ 1,500/mm3 Plt ≥ 100,000/mm3 Hb ≥ 9 g/dL (may have had blood transfusions) AST/ALT ≤ 2.5 IULN or ≤ 5 IULN with known liver metastases Total bilirubin ≤ 1.5 IULN Serum Creatinine ≤ 1.5 IULN INR ≤ 1.5 and PTT ≤ 1.5 IULN

Exclusion Criteria:

* Previous exposure to an anti-EGFR therapy or irinotecan-based chemotherapy
* Radiotherapy, surgery (excluding previous diagnostic biopsy), or any investigational drug in the 30-day period before the start of treatment in our trial
* Female patients who are pregnant or lactating
* Patients with any history of another primary malignancy in the past five years, with the exception of non-melanoma skin cancer, and carcinoma in situ of uterine cervix
* Patients with history of allergic reactions attributed to compounds of similar chemical or biologic drugs as cetuximab, irinotecan, fluorouracil or leucovorin
* Adjuvant treatment that was terminated 6 months or less before the start of treatment in our trial
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | PFS was measured from the start of chemotherapy to the date of disease progression or to the date of death if no progression whichever came first, assessed up to 26 weeks
  PFS is defined as the time from the date of randomization to the first date of documentation progression (per investigator assessment) or death as a result of any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | 26 weeks after study start
  Overall survival OS is defines as the time from date of randomization to date of death due to any cause
Objective Response rate | 26 weeks after study start
  Tumor response was defined as partial and complete responses, according to the RECIST criteria.
Time of treatment failures | 26 weeks after study start
  Time of treatment failures define as the time from the date of randomization to the date of each of the following,
  * The treatment modalities did not destroy or modify the cancer cell.
  * The tumor either became larger (disease progression) or stayed the same size after treatment,
  * Death from any cause
  * Discontinuation of treatment
Adverse events | 26 weeks after study start
  Safety wills assess on the basis of reports of adverse events, laboratory-test results, and vital sign measurements. Adverse events were categorized According to the Common Toxicity Criteria of the National Cancer Institute, version 4.0, in which a grade of 1 indicates mild adverse events, a grade of 2 moderate adverse events, a grade of 3 serious adverse events, and a grade of 4 life-threatening adverse events
immunogenicity | 26 weeks after study start
  antidrug antibody [ADA] and neutralizing antibody [nAb] assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Taleqani Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided